CLINICAL TRIAL: NCT04381780
Title: Treatment of Fibromyalgia With a Unique Polypeptide Nutritional Support
Brief Title: Treatment of Fibromyalgia With Recovery Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Practitioners Alliance Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN Study RF-2- 2020
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: Open pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessing clinical outcomes (Experimental): Nutritional support with Recovery Factors
  Interventions: Dietary Supplement: Recovery Factors

INTERVENTIONS:
Dietary Supplement: Recovery Factors — A unique porcine serum based polypeptide nutritional support

SUMMARY:
Treatment of Fibromyalgia and CFS with Recovery Factors

DETAILED DESCRIPTION:
Use of a unique oral porcine peptide nutritional supplement in those meeting ACR 2010(amended) diagnostic criteria for Fibromyalgia or CDC Criteria for CFS

ELIGIBILITY:
Inclusion Criteria:

* Meet the ACR 2010 Amended Fibromyalgia Diagnostic Criteria or CFS CDC criteria; Score 5 or less on Energy VAS

Exclusion Criteria:

Under 18 Pregnant Other severe complicating conditions

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Composite VAS | 6 weeks
  Composite of VAS for Fatigue, sleep, cognition, pain and overall well being

SECONDARY OUTCOMES:
FIQ-R | 1 month
  Fibromyalgia Impact Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Jacob Teitelbaum MD, Kailua, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No